CLINICAL TRIAL: NCT06827041
Title: Use of Phage Therapy for Treatment of a Life-Threatening, Multidrug Resistant Staphylococcus Epidermidis Chronic Periprosthetic Joint Infection: an N-of-1 Trial
Brief Title: Use of Phage Therapy for Treatment of a Periprosthetic Joint Infection
Acronym: BPhage
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Cytophage Technologies Inc. (Unknown)
Responsible Party: Principal Investigator, Marisa Azad, Assistant Professor of Medicine, Ottawa Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20231130
Record Dates: First submitted 2024-04-03; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Periprosthetic Joint Infection

STUDY DESIGN:
Intervention Model Description: Lytic monophage prepared in injection-grade saline will be given via two routes:
  1. intravenously twice daily, and concomitantly,
  2. intraarticularly twice daily, for a total duration of 14 days. In addition to phage therapy, the patient will receive standard of care antibiotic therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phage therapy (Experimental): Lytic monophage prepared in injection-grade saline will be given via two routes: a) intravenously twice daily, and concomitantly, b) intra-articularly twice daily, for a total duration of 14 days. In addition to phage therapy, the patient will receive standard of care antibiotic therapy.
  Interventions: Biological: Phage (Cytophage Technologies)

INTERVENTIONS:
Biological: Phage (Cytophage Technologies) — Our phage is a new type of investigational treatment for bacterial infections. Our lytic, monophage preparation was provided by Cytophage Technologies and underwent rigorous testing to ensure final product potency (7 x 10^9 PFU/dose), purity, fidelity, and safety; laboratory tests demonstrate phage in vitro efficacy against the S. epidermidis strain.
  Phage prepared in injection-grade saline will be given via two routes: a) intravenously twice daily, and concomitantly, b) intraarticularly twice daily, for a total duration of 14 days.

SUMMARY:
The goal of this clinical trial is to learn about the safety, tolerability and activity or efficacy of systemic intravenous and intraarticular administration of a mono-bacteriophage (phage) peparation in a patient with chronic-recalcitrant methicillin-resistant Staphylococcus epidermidis (MRSE) periprosthetic joint infection (PJI) and also to understand clinical changes pre- and post-therapy, as well as identifying adjunctive changes in biomarkers (C-reactive protein [CRP], erythrocyte sedimentation rate [ESR], and interleukin-6 [IL-6]) correlated with PJI.

Phage will be administered to the study participant with chronic PJI twice daily over a total duration of two weeks via two routes: a) intravenous (through vein) and b) intra-articular (through the affected joint). Phage therapy is given 4 hours after the patient receives their standard of care antibiotic therapy. The patient will remain in clinical follow-up for up to a year.1

DETAILED DESCRIPTION:
At The Ottawa Hospital (TOH), the orthopedic infectious diseases team is currently managing a very challenging case: a 78-year-old female with a severe, chronic-recalcitrant right hip PJI due to a multidrug resistant strain of S. epidermidis in which surgical source control with complete removal of implants cannot be achieved, and in whom there are no viable antibiotic treatment options for chronic suppressive therapy. This patient has undergone multiple surgical revisions with complex reconstructions and adjunctive flap coverage procedures and has received prolonged courses of antibiotic therapy. Unfortunately, this patient suffered multiple, severe antibiotic allergic reactions during initial treatment course which has precluded the use of any viable suppressive therapy - a treatment strategy which is critical to preventing relapse of infection and is at the crux of chronic PJI management.

In the absence of any viable adjunctive antimicrobial therapy, this patient is at very high risk of mortality. The Investigators have exhausted all surgical and medical management of PJI for our patient. Remaining on lower dose daptomycin and adjunctive oral rifampin, the patient continued to experience myalgias and neuropathy. It was anticipated that with eventual discontinuation of daptomycin (this patient cannot remain indefinitely on this therapy given her symptoms), her infection would again rapidly relapse with systemic symptoms. This infection is associated with a high risk of mortality without a viable suppressive antimicrobial treatment; a more aggressive surgical approach (high right leg amputation and hemipelvectomy) to reduce the burden of infection is not possible in this patient given her frailty, co-morbidity, resultant significant physical debility and risk of surgical complications. Given the above, phage therapy poses very low risk and is a remaining possible medical therapy that may eradicate her infection.

The primary objective of this study is to investigate the safety, tolerability and activity or efficacy of systemic (intravenous) and intra-articular administration of phage in our patient with chronic-recalcitrant methicillin-resistant S. epidermidis PJI.

Secondary objectives will be documenting clinical changes pre- and post-therapy, as well as identifying adjunctive changes in biomarkers (C-reactive protein [CRP], erythrocyte sedimentation rate [ESR], and interleukin-6 [IL-6]) correlated with PJI.

In this study, lytic phage prepared in injection-grade saline will be administered to the patient both intravenously and intraarticularly, twice a day for a duration of 14 days. In addition to phage therapy, the patient will receive standard of care antibiotic therapy.

The patient will remain in clinical follow-up for up to one year.

ELIGIBILITY:
Inclusion Criteria:

This N-of-1 Phage therapy is designed for one patient who meet the following conditions.

* willingness to provide signed and dated informed consent form to participate in the clinical study.
* severe chronic periprosthetic joint infection due to a multidrug resistant strain of S. epidermidis in which surgical source control with complete removal of implants cannot be safely achieved
* have received multiple surgical revisions with complex reconstructions and adjunctive flap coverage procedures and prolonged courses of antibiotic therapy and suffered multiple, severe antibiotic allergic reactions during initial treatment course which has lead to the use of any viable suppressive therapy impossible
* complex burden of hardware
* poor bone quality and hip instability with high associated morbidity and mortality due to the S. epidermidis infection

Exclusion Criteria:

- below age 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Safety of phage therapy | From first day to 12 months from treatment
  Reactions and adverse events to study treatment.
Efficacy of phage therapy (clinical response) | 1 year
  Wound healing and no recurrence of the infection as determined by the orthopedic infectious diseases physician during follow-up to 12 months from phage treatment.

SECONDARY OUTCOMES:
Response of laboratory markers (C-reactive protein) of inflammation to phage treatment | 1 year
  Serum C-reactive protein (mg/L) as measured at baseline, during phage treatment to day 14, and in follow-up to 12 months from phage treatment.
Response of laboratory markers (erythrocyte sedimentation rate) of inflammation to phage treatment | 1 year
  Serum erythrocyte sedimentation rate (mm/hr) as measured at baseline, during phage treatment to day 14, and in follow-up to 12 months from phage treatment.
Response of laboratory markers (peripheral blood neutrophil count) of inflammation to phage treatment | 1 year
  Peripheral blood neutrophil count (cells/L) as measured at baseline, during phage treatment to day 14, and in follow-up to 12 months from phage treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa A Azad, MD PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available from a publication which is pending
Supporting Information: CSR
Time Frame: 12 months from study treatment
Access Criteria: Any desired information may be requested directly of the principal investigator